CLINICAL TRIAL: NCT07399912
Title: Engaging Home-monitored Assessment to Navigate Clinical Decision-making -The ENHANCe Study
Brief Title: Engaging Home-monitored Assessment to Navigate Clinical Decision-making
Acronym: ENHANCe
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: SingHealth Polyclinics (Other)
Collaborators: Nanyang Polytechnic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2024-4269-APP1
Record Dates: First submitted 2025-12-28; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-09

CONDITIONS: Hypertension,Essential
Keywords: Hypertension; Home blood pressure; Primary Care; Clinical decision support system
MeSH Terms: conditions — Essential Hypertension; Hypertension | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Parallel Cluster RCT
Who Masked: Participant
Masking Description: Patient Participants will be blinded to the group they are allocated to
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypertension management using the Clinical Decision Support System (Experimental): All patients will have access to online educational resources throughout the study. After recruitment, they will receive a nurse-led education on HBP monitoring. The research team will train all primary care physicians (PCPs) on managing patients with hypertension using HBP records. The PCPs in the intervention group will be briefed on how the ENHANCe app works, and its recommendations. The ENHANCe app will be installed on designated mobile phones, and research staff will analyse HBP records during visits, documenting the output for PCPs to use. Based on the app's recommendations, patients will consult with intervention group PCPs 2-3 times throughout the study, with the last follow-up at 6 months. PCPs will complete a consult checklist after each visit. FGDs will be conducted with PCPs at the end of the study. The interviews will be recorded and transcribed for analysis.
  Interventions: Device: ENHANCe app; Other: Teaching and training
- Hypertension management as per usual care without a clinical decision support system (Other): All patients will have access to online educational resources throughout the study. After recruitment, they will receive a nurse-led education on HBP monitoring. The research team will train all primary care physicians (PCPs) on managing patients with hypertension using HBP records. Control group PCPs will manage patients using HBP records at their discretion, with a final follow-up scheduled at 6 months. PCPs will complete a consult checklist after each visit. Research staff will use the ENHANCe app to analyse BP diaries and document outcomes, but control group PCPs will not have access to the app or its results.
  Interventions: Other: Teaching and training; Other: Usual care

INTERVENTIONS:
Device: ENHANCe app — ENHANCe app is a prototype; it is a smartphone based clinical decision support (CDS) tool to manage patients with hypertension using their home blood pressure. The app will scan patients' home BP records from paper or mobile phone, and provide a recommendation to the doctor on how to manage their blood pressure. The patient will not need to use the device during the study period. However, the recommendation from the ENHANCe app will be available to the doctor to manage your blood pressure during the study period if the patient is in the intervention group.
  Arms: Hypertension management using the Clinical Decision Support System
Other: Teaching and training — All patients will have access to online educational resources throughout the study. After recruitment, they will receive a nurse-led education on HBP monitoring. The research team will train all primary care physicians (PCPs) on managing patients with hypertension using HBP records.
Other: Usual care — Physicians manage patients using HBP records at their discretion
  Arms: Hypertension management as per usual care without a clinical decision support system

SUMMARY:
This study is testing a new app called ENHANCe, which is designed to help family doctors manage patients with high blood pressure using readings taken at home.

DETAILED DESCRIPTION:
The researchers want to find out if the app is easy to use in everyday clinic settings, whether doctors find it helpful and are willing to use it, and if it helps improve care. The study will involve 16 doctors and 100 patients with high blood pressure, split into two groups at two clinics. One group will use the ENHANCe app, which can read blood pressure data from different sources-including handwritten notes-and give doctors advice based on that information. The other group will receive regular care without the app. Over six months, researchers will collect feedback from doctors through surveys and group discussions at the end of the study. They'll also track how many people complete the study, how long clinic visits take, whether doctors follow the app's advice, and how well patients' blood pressure is controlled. The goal is to see if the app can help doctors make faster, better decisions and improve health outcomes for people managing their blood pressure at home.

ELIGIBILITY:
Inclusion Criteria:

For primary care physicians:

* PCPs aged 21 years and above.
* Involved in the clinical management of patients with hypertension in the past six months.

For patients:

* Patients aged 21 years and above
* Documentation of hypertension diagnosis in EMR
* Owns an HBP monitoring device

Exclusion Criteria for patients:

* Documentation of dementia diagnosis in EMR
* Audio or visual impairments
* Hypertensive urgency or emergency

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Response rate of participants | 6 months
  Participants agreeable to participate in the study
Agreement with the CDSS recommendation among PCPs | 6 months
  Proportion of PCPs who agree with the CDSS recommendation in the two groups
Withdrawal rate | 6 months
  Proportion of participants who withdrew
Study completion rate | 6 months
  Proportion of participants who completed the intervention
Adverse event rates | 6 months
  Proportion of adverse events reported in the two groups
Consult duration | 6 months
  Consult time in the groups
Ease of home blood pressure record assessment among PCPS | 6 months
  Ease of home blood pressure record assessment among PCPS in the two arms

SECONDARY OUTCOMES:
Proportion of CDSS recommendation followed by the PCPS | 6 months
  Proportion of ENHANCe recommendations followed by the PCPs among the two groups
Blood pressure control status | 6 months
  Blood pressure control status among patients in the two groups

CONTACTS AND LOCATIONS:
Locations (1):
- SingHealth Polyclinics, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared